CLINICAL TRIAL: NCT03484299
Title: Chemotherapy and Irreversible Electroporation (IRE) in the Treatment of Advanced Pancreatic Adenocarcinoma
Brief Title: Chemotherapy and Irreversible Electroporation in the Treatment of Advanced Pancreatic Adenocarcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Robert C. Martin, Principal Investigator, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17.0529
Record Dates: First submitted 2018-02-13; First posted 2018-03-30 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Electroporation; Gemcitabine; folfirinox

STUDY DESIGN:
Intervention Model Description: All subjects undergoing IRE will receive treatment with either FOLFIRINOX or gemcitabine (based on which regimen was received prior to IRE)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Other): Irreversible electroporation and treatment with either FOLFIRINOX or Gemcitabine (based upon which chemotherapy regimen received prior to IRE)
  Interventions: Procedure: Irreversible Electroporation (IRE); Drug: Gemcitabine; Drug: FOLFIRINOX

INTERVENTIONS:
Procedure: Irreversible Electroporation (IRE) — Non-thermal ablation of tumor
Drug: Gemcitabine — 25% dose - first 3 enrolled; 50% dose - next 3 enrolled; 75% dose - remaining 4 enrolled
Drug: FOLFIRINOX — 25% dose - first 3 enrolled; 50% dose - next 3 enrolled; 75% dose - remaining 4 enrolled

SUMMARY:
Compare the efficacy and tolerability of IRE in combination with either FOLFIRINOX or gemcitabine in patients with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
Phase II study in which all patients undergoing IRE for the treatment of locally advanced pancreatic carcinoma will receive either FOLFIRINOX or gemcitabine as peri-ablation treatment.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 18 years of age
* diagnosed with stage III pancreatic cancer
* tumor is measurable
* GFR > mL/min/1.73m2
* willing and able to comply with protocol requirements
* AST/ALT >3 times upper limit of normal
* stable surgical post-operative course as defined by operative surgeon

Exclusion Criteria:

* participating in another clinical trial for the treatment of cancer at the time of screening
* pregnant or currently breast feeding
* have a cardiac pacemaker or ICD implanted that cannot be deactivated during IRE procedure
* have non-removable implants with metal parts within 1 cm of the target lesion
* had a myocardial infarction within 3 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-30 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse and Serious Adverse events will be captured (safety and tolerability) | Time from first dose until subject has reached 90 days post last active study treatment
  Adverse and Serious Adverse events will be collected and analyzed

SECONDARY OUTCOMES:
Progression free survival | Time from first dose date to first date of confirmed disease progression, assessed for 90 days
  Triphase CT scan will be performed within one month of IRE procedure. Triphase CT scans will then be obtained every 3 months to check disease status.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Martin, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Bhutiani N, Li Y, Zheng Q, Pandit H, Shi X, Chen Y, Yu Y, Pulliam ZR, Tan M, Martin RCG 2nd. Electrochemotherapy with Irreversible Electroporation and FOLFIRINOX Improves Survival in Murine Models of Pancreatic Adenocarcinoma. Ann Surg Oncol. 2020 Oct;27(11):4348-4359. doi: 10.1245/s10434-020-08782-2. Epub 2020 Jul 17. PMID 32681477